CLINICAL TRIAL: NCT01179308
Title: The Effect of Adding Intraoperative Regional Anesthesia on Cancer Recurrence in Patients Undergoing Lung Cancer Resection
Brief Title: Regional Anesthesia and Lung Cancer Recurrence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator decided to close this study site.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Andrea Kurz, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10-610; NCT00999726 (obsolete NCT alias)
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Lung Cancer
Keywords: regional analgesia; routine general anesthesia; immune system response; lung cancer (stage 1-3)
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- General-epidural anesthesia (Active Comparator): Epidural and general anesthesia
  Interventions: Other: General-epidural anesthesia
- General anesthesia (Active Comparator): General anesthesia alone
  Interventions: Other: Balanced general anesthesia and postoperative opioids

INTERVENTIONS:
Other: General-epidural anesthesia — General anesthesia combined with epidural anesthesia
  Arms: General-epidural anesthesia
Other: Balanced general anesthesia and postoperative opioids — General anesthesia alone
  Arms: General anesthesia

SUMMARY:
Test the effect of combined regiona/general anesthesia on lung cancer recurrence compared to general anesthesia alone.

DETAILED DESCRIPTION:
Surgery is the primary treatment of lung cancer, but surgery releases tumor cells into the systemic circulation. Whether this minimal residual disease results in clinical metastases is a function of host defense. At least three perioperative factors shift the balance toward initiation and progression of minimal residual disease. (1) Surgery per se depresses cell-mediated immunity, reduces concentrations of tumor-related anti-angiogenic factors (e.g., angiostatin and endostatin), and increases concentrations of pro-angiogenic factors such as VEGF. (2) Anesthesia impairs numerous immune functions, including neutrophil, macrophages, dendritic cells, T lymphocytes (T-cell), and Natural killer cell (NK-cell) functions. (3) Opioid analgesics inhibit both cellular and humoral immune function in humans, and promote tumor growth in rodents. Regional analgesia attenuates each of these adverse effects. For example, regional anesthesia largely prevents the neuroendocrine stress response to surgery by blocking afferent neural transmission. With combined regional and general anesthesia/analgesia, the amount of general anesthetic required is much reduced - as is, presumably, immune suppression. And finally, regional analgesia provides superb pain relief, essentially obliterating the need for postoperative opioids. Animal studies show that regional anesthesia improves natural kill cell function and reduces the metastatic burden in animals inoculated with carcinoma cells. Preliminary retrospective data in cancer patients showed, that paravertebral analgesia for breast cancer surgery reduced risk of recurrence or metastasis by 40% during a 2.5 to 4-year follow-up period.

The investigators thus propose to evaluate the effect of combined epidural-general anesthesia compared to general anesthesia on cancer recurrence semi-annually over a period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary non-small cell lung cancer (stage 1-3) as determined according to the IASLC Lung Cancer Staging Project;
* Scheduled for potentially curative tumor resection;
* Written informed consent, including willingness to be randomized to epidural anesthesia/analgesia plus general anesthesia or to general anesthesia and postoperative opioid analgesia.

Exclusion Criteria:

* Any contraindication to epidural anesthesia, (including coagulopathy, abnormal anatomy).
* Any contraindication to midazolam, propofol, sevoflurane, fentanyl, morphine, or hydromorphone.
* Age < 18 or > 85 years old.
* Other cancer not believed by the attending surgeon to be in long-term remission.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
disease-free survival | up to 5 years after surgery
  The effect of regional versus general anesthesia on the primary outcome of disease-free survival (time to the earlier or recurrence or death from any cause)

SECONDARY OUTCOMES:
NK cell function | up to three years post procedure
  Secondary outcomes measured at repeated perioperative time points, include NK cell function, immune-function markers (cytokines, cortisol) and pain.
Immune function markers | for up to 3 years post procedure
  Secondary outcomes measured at repeated perioperative time points, include NK cell function, immune-function markers (cytokines, cortisol) and pain.
Pain | up to 3 years post proceudure
  Secondary outcomes measured at repeated perioperative time points, include NK cell function, immune-function markers (cytokines, cortisol) and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, M.D., Principal Investigator — The Cleveland Clinic
Locations (2):
- Cleveland Clinic, Cleveland, Ohio, United States
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No